CLINICAL TRIAL: NCT06934720
Title: Active Physical Activity - Virtual Reality Cognitive Therapy
Brief Title: VR-based Physical Activity and Reminiscence Therapy
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hong Kong University of Science and Technology (Other)
Responsible Party: Principal Investigator, GE LIN KAN, Professor, Hong Kong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HREP20220139; FS110 (Other Grant/Funding Number: Hong Kong University of Science and Technology)
Record Dates: First submitted 2025-04-05; First posted 2025-04-18 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Dementia; Neurodegenerative Disease; Mild Cognitive Impairment (MCI); Virtual Reality; Physical Activity; Alzheimer's Disease (AD); Cognitive Therapy
MeSH Terms: conditions — Dementia; Neurodegenerative Diseases; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial: Eligible participants will be randomly assigned to either the intervention or control group. Each participant will attend sessions at least twice weekly (15-30 minutes per session) over 12 weeks.
  Given the setting in nursing homes, variability in health status and potential hospitalizations will be accounted for. An additional three weeks will be allowed for compensatory sessions, resulting in a total duration of 12-15 weeks.
  Participants may stop or drop out of the study at any time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Behavioral: aPAVRCT
- control (No Intervention): usual care (PA)

INTERVENTIONS:
Behavioral: aPAVRCT — * We offered a system integrated with an indoor bike (for physical activity) and a multisensory VR environment (for cognitive training, such as reminiscence).
  * Participants will actively navigate the virtual environment by pedaling and steering the handlebar.
  * Care professionals will deliver the intervention using this system.
  Arms: Experimental

SUMMARY:
The goal of this clinical trial is to learn if active Physical activity + virtual reality cognitive therapy (aPAVRCT) works to slow the progression of AD cognitive decline in older adults. It will also learn about the physical effects and mental effects of the aPAVRCT. The main questions it aims to answer are:

Does aPAVRCT slow the progression of AD cognitive decline? (e.g., HK-MoCA, ADAS-Cog) Does aPAVRCT improve physical function? (e.g., ADL) Does aPAVRCT improve mental health? (e.g., GDS-15, PANAS) Does aPAVRCT improve life satisfaction? Does aPAVRCT improve other cognitive or physical capacities? What issues and benefits do participants and stakeholders (e.g., families, caregivers, managers) have when taking aPAVRCT? (e.g., NPI-Q) Researchers will compare the intervention group (aPAVRCT) to a control group (rehabilitation bike) to see if aPAVRCT works to slow the progression of AD in cognitive decline.

Participants will:

Take aPAVRCT (interventional group) or usual physical acitvity (control group) at least twice a week, 15 minutes for each session, for 12-16 weeks Physiotherapies (assistants) and care professionals will do the intervention, research group will operate, observe, and assist the experiment.

All the experiment processes will be recorded. Visit the sites everyday for checkups and tests Keep a diary of their symptoms, the number of times, and any essential information

Sites: around 3-5 nursing homes, under one institution. Inclusion criteria: older adults in the setting who have the ability to pedal a rehabilitation bike.

DETAILED DESCRIPTION:
The aim of study is to investigate the effect of active Physical activity + virtual reality cognitive therapy (aPAVRCT) on cognitive function in older adults with Alzheimer's Dementia and related dementias. The investigator hypothesizes the "Physical activity + virtual environment brain stimulations' would slow the process of AD cognitive decline. The life satisfaction score in the intervention group would be higher than that of the control group.

The investigator will conduct measurements on three aspects: The Chinese version of the MoCA, physical functions, and emotional changes. Data will be collected at baseline, 4-week, 8-week, 12-week after interventions for the two groups, and a follow-up measurement. In addition, the investigator will use some qualitative methods, such as focus group, interview, observation, during and after the first 3-month intervention to identify some issues during the intervention and to probe caregivers. The investigator will use both the Ttest between the two groups (to compare cognitive decline progressions, and life satisfaction) and mixed methods to illustrate life satisfaction, especially among caregivers.

ELIGIBILITY:
Inclusion Criteria:

* older adults in the setting who have the ability to pedal the rehabilitation bike

Exclusion Criteria:

* Individuals self-reporting or identified by stakeholders as unwilling or unsuitable to participate.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-19 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Hong Kong - Montreal cognitive assessment scale | at the baseline, during intervention (4-week, 8-week, 12-week, 16-week), and post-intervention assessment (3 months, 6 months after the intervention)
  MoCA is a cognitive assessment method for dementia, particularly mild stages of cognitive impairment. (range, 0-30, with lower scores indicating greater cognitive impairment)
The Integrated Alzheimer's Disease Rating Scale (iADRS) | at the baseline, during intervention (4-week, 8-week, 12-week, 16-week), and post-intervention assessment (3 months, 6 months after the intervention)
  iADRS (range, 0-144, with lower scores indicating greater cognitive and functional described impairment) is to assess both cognitive and physical functions for dementia, combines the 13-item cognitive subscale of the Alzheimer's Disease Assessment Scale (ADAS-Cog13 ), the Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living Inventory (ADCS-iADL).
Mini-Mental State Examination (MMSE) | at the baseline, during intervention (4-week, 8-week, 12-week, 16-week), and post-intervention assessment (3 months, 6 months after the intervention)
  For cognitive assessment, (range: 0-144, with lower scores indicating greater cognitive impairment)

SECONDARY OUTCOMES:
Time up and Go Test | at the baseline, during intervention (4-week, 8-week, 12-week, 16-week), and post-intervention assessment (3 months, 6 months after the intervention)
  TUG test evaluates fall risk, mobility and physical performance in the elderly
Sit to Stand Test | at the baseline, during intervention (4-week, 8-week, 12-week, 16-week), and post-intervention assessment (3 months, 6 months after the intervention)
  sit to stand test is a test that evaluates the functional strength of the lower extremity, balance and fall risk.
Geriatric depression scale (GDS-15) | at the baseline, during intervention (4-week, 8-week, 12-week, 16-week), and post-intervention assessment (3 months, 6 months after the intervention)
  Geriatric depression scale identifies possible depression in older adults. Range: 0-15, with higher scores indicating greater possible depression.
The Cornell Scale for Depression in Dementia (CSDD) | at the baseline, during intervention (4-week, 8-week, 12-week, 16-week), and post-intervention assessment (3 months, 6 months after the intervention)
  CSDD is to assess changes in a person's mood, behaviours and routines which may be symptoms of depression. Range: 0-38, with higher scores indicating greater depression symptoms
Neuropsychiatric Inventory-Questionnaire (NPI-Q) | at the baseline, during intervention (4-week, 8-week, 12-week, 16-week), and post-intervention assessment (3 months, 6 months after the intervention)
  NPI-Q is to interview informant for symptom severity and caregiver distress. Range: 0-36, higher score indicates greater neuropsychiatric disturbances or caregiver distress.
Positive Affect and Negative Affect Scale | at the baseline, during intervention (4-week, 8-week, 12-week, 16-week), and post-intervention assessment (3 months, 6 months after the intervention)
  PANAS is used to assess positive and negative emotional status and changes. This self-report questionnaire consists of two 10-item scales to measure positive and negative. The total score is calculated by finding the sum of the 10 positive items, and then the 10 negative items. Scores range from 10 - 50 for both sets of items. For the total positive score, a higher score indicates more of a positive affect. For the total negative score, a lower score indicates less of a negative affect.